CLINICAL TRIAL: NCT07074548
Title: The Effect of Hydroxytyrosol on Improving Neutrophil-to-Lymphocyte Ratio, Monocyte-to-Lymphocyte Ratio, and Superoxide Dismutase in Pregnant Women With Hypertension: A Randomized Controlled Trial
Brief Title: Effect of Hydroxytyrosol on NLR, MLR, and SOD in Hypertensive Pregnant Women
Acronym: HyPreg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Damar Prasmusinto, Consultant Maternal-Fetal Medicine Specialist, ObstetricianGynecologist and Principal Investigator, Dr Cipto Mangunkusumo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25-03-0308
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Hypertension in Pregnancy
Keywords: hydroxytyrosol
MeSH Terms: conditions — Hypertension, Pregnancy-Induced | interventions — 3,4-dihydroxyphenylethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study uses identical capsules for hydroxytyrosol and placebo to maintain masking of all parties.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): Participants in this arm will receive a placebo capsule orally once daily for 4 weeks, alongside standard antenatal care. The placebo is visually identical to the hydroxytyrosol supplement to maintain masking.
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Hydroxytyrosol
- Hydroxytyrosol Group (Active Comparator): Participants in this arm will receive hydroxytyrosol 10 mg orally once daily for 4 weeks, alongside standard antenatal care.
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Hydroxytyrosol

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo oral capsule identical in appearance to hydroxytyrosol supplement, administered once daily for 4 weeks.
Dietary Supplement: Hydroxytyrosol — Hydroxytyrosol is a natural polyphenol with antioxidant and anti-inflammatory properties, derived from olives. In this study, hydroxytyrosol 10 mg will be administered orally once daily for 4 weeks to assess its effects on blood pressure and inflammatory biomarkers in hypertensive pregnant women.

SUMMARY:
The goal of this clinical trial is to evaluate whether hydroxytyrosol supplementation (10 mg/day for 4 weeks) is effective in improving inflammatory and oxidative stress markers in pregnant women diagnosed with hypertensive disorders of pregnancy (including preeclampsia, chronic hypertension, and gestational hypertension). The main questions it aims to answer are:

1. Does hydroxytyrosol supplementation reduce neutrophil-to-lymphocyte ratio (NLR) and monocyte-to-lymphocyte ratio (MLR)?
2. Does hydroxytyrosol supplementation lower systolic and/or diastolic blood pressure?
3. Does hydroxytyrosol supplementation increase superoxide dismutase (SOD) levels?

Researchers will compare a group receiving hydroxytyrosol supplementation to a standard care control group to see if hydroxytyrosol produces superior anti-inflammatory and antioxidant effects.

Participants will:

* Take hydroxytyrosol 10 mg orally once daily for 4 weeks (intervention group) or receive standard antenatal care without hydroxytyrosol (control group).
* Undergo laboratory testing (NLR, MLR, SOD) before and after the intervention.
* Have their blood pressure monitored regularly throughout the study period.

DETAILED DESCRIPTION:
Hypertensive disorders of pregnancy, including preeclampsia, chronic hypertension, and gestational hypertension, are major contributors to maternal and perinatal morbidity and mortality worldwide. Oxidative stress and systemic inflammation play critical roles in the pathophysiology of HDP. Biomarkers such as the neutrophil-to-lymphocyte ratio (NLR), monocyte-to-lymphocyte ratio (MLR), and superoxide dismutase (SOD) have been associated with the severity and progression of these conditions.

Hydroxytyrosol, a polyphenol compound found in olives, has demonstrated potent antioxidant and anti-inflammatory properties in both in vitro and in vivo studies. Its potential therapeutic role in cardiovascular and metabolic diseases suggests a possible benefit in hypertensive pregnancies, though clinical evidence in this population remains limited.

This randomized controlled trial aims to evaluate the effectiveness of hydroxytyrosol supplementation (10 mg/day for 4 weeks) in improving markers of systemic inflammation and oxidative stress among pregnant women with HDP. A total of eligible pregnant women diagnosed with preeclampsia, chronic hypertension, or gestational hypertension will be randomly assigned to receive either hydroxytyrosol supplementation in addition to standard antenatal care (intervention group), or standard antenatal care alone (control group).

The primary outcome measures include changes in NLR and MLR after 4 weeks of supplementation. Secondary outcomes include changes in systolic and diastolic blood pressure, NLR and MLR levels, and serum SOD levels. All participants will undergo baseline and post-intervention laboratory testing and blood pressure monitoring.

The results of this study are expected to provide clinical insight into the potential role of hydroxytyrosol as a supportive therapeutic agent in managing hypertensive disorders during pregnancy, potentially improving maternal outcomes through modulation of oxidative stress and inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy with a live intrauterine fetus
2. Gestational age over 24 weeks. Gestational age is confirmed based on:

   * Last Menstrual Period (LMP)
   * First trimester ultrasound biometry
3. Belongs to the Hypertensive Disorders of Pregnancy group, with the following criteria:

   * Gestational hypertension and preeclampsia according to ACOG 2018 criteria
   * Chronic hypertension according to ACOG 2019 criteria
   * Superimposed preeclampsia according to ACOG 2018 criteria

Exclusion Criteria:

1. Pregnancy with infection, including chronic infections such as tuberculosis (TB), HIV, or hepatitis B
2. Pregnancy with other complications (e.g., diabetes mellitus, heart disease, kidney disease, liver disease, malignancy, autoimmune disorders)
3. Refusal to participate in the study

Ages: 24 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 42 (Actual)
Dates: Start 2025-07-10 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Neutrophil-to-Lymphocyte Ratio (NLR), MLR (Monocyte-to-Lymphocyte Ratio), and SOD (Superoxide Dismutase level) from Baseline to Week 4 | Baseline and Week 4
  To evaluate the anti-inflammatory effect of hydroxytyrosol supplementation by comparing the change in NLR, MLR, SOD levels between the hydroxytyrosol and placebo groups after 4 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Cipto Mangunkusumo National Central Public Hospital, Jakarta Pusat, Jakarta Special Capital Region, Indonesia